CLINICAL TRIAL: NCT01990339
Title: Takepron Specified Drug-use Survey "Gastroesophageal Reflux Disease With Dyspepsia Symptoms"
Brief Title: Lansoprazole Tablets Special Drug Use Surveillance Gastroesophageal Reflux Disease With Dyspepsia Symptoms
Acronym: LEGEND
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 467-531; JapicCTI-132310 (Registry Identifier: Japic CTI); JapicCTI-R140645 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Gastroesophageal Reflux Disease With Dyspepsia Symptoms
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lansoprazole: Lansoprazole (Takepron), tablets, orally, once daily for up to 8 weeks. Reflux esophagitis: the usual adult dosage is 30 mg of lansoprazole. For maintenance therapy of repeatedly recurring/relapsing reflux esophagitis, the dosage is 15 mg of lansoprazole administered orally once daily. If insufficient efficacy is observed, the dosage may be increased to 30 mg administered orally once daily. Nonerosive gastroesophageal reflux disease: the usual adult dosage is 15 mg of lansoprazole administered orally once daily for up to 4 weeks.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — • Reflux esophagitis The usual adult dosage is 30 mg of lansoprazole administered orally once daily for up to 8 weeks.
  For maintenance therapy of repeatedly recurring/relapsing reflux esophagitis, the dosage is 15 mg of lansoprazole administered orally once daily. If insufficient efficacy is observed, the dosage may be increased to 30 mg administered orally once daily.
  • Nonerosive gastroesophageal reflux disease Non-erosive gastroesophageal reflux disease The usual adult dosage is 15 mg of lansoprazole administered orally once daily for up to 4 weeks.
  Other Names: Takepron

SUMMARY:
To evaluate the efficacy of 4-week lansoprazole (Takepron) therapy for subjective symptomatic improvement in gastroesophageal reflux disease patients with dyspepsia symptoms

DETAILED DESCRIPTION:
This is a special drug use surveillance of lansoprazole (Takepron) with a 4-week observational period, designed to evaluate the efficacy in gastroesophageal reflux disease patients with dyspepsia symptoms (planned sample size, 15000).

The dosage regimen is as follows:

* For reflux esophagitis, the usual adult dosage is 30 mg of lansoprazole administered orally once daily for up to 8 weeks. For maintenance treatment of repeatedly recurring/relapsing reflux esophagitis, the dosage is 15 mg of lansoprazole administered orally once daily. If insufficient efficacy is observed, the dosage may be increased to 30 mg administered orally once daily.
* For non-erosive gastroesophageal reflux disease, the usual adult dosage is 15 mg of lansoprazole administered orally once daily for up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with heartburn or acid regurgitation at the start of Takepron administration* , or patients without heartburn and acid regurgitation, but with endoscopic findings classified as Los Angeles grade A-D at the start of Takepron therapy.
2. Patients with symptoms of dyspepsia (i.e., postprandial fullness, early satiation, epigastric pain, epigastric burning, upper abdominal bloating, nausea/vomiting, or belching) at the start of Takepron administration* *These patients must have answered "never, " "sometimes/mild," "often/moderate," or "frequent/severe" on a 4-point scale questionnaire about subjective symptoms.

Exclusion Criteria:

1. Patients who have taken any proton pump inhibitors (including Takepron) within 4 weeks before the start of Takepron administration
2. Patients taking antidepressants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastroesophageal reflux disease with dyspepsia symptoms
Sampling Method: Non-Probability Sample
Enrollment: 14965 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study during the period between December 8, 2008 and June 30, 2010.
Pre-assignment Details: Participants enrolled in the study were clinically diagnosed with reflux esophagitis or non-erosive gastroesophageal reflux disease.
Period: Overall Study
Arm/Group | Lansoprazole
Started | 14965
Completed | 12653
Not Completed | 2312
Not completed — Data Not Available | 49
Not completed — Voluntary Withdrawal | 1402
Not completed — Lost to Follow-up | 861

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set included all enrolled participants with data available (8 patents were excluded for medical reasons; 41 were excluded for other reasons), 1402 patients who did not visit the study site after initial prescription and 861 patients whose questionnaires were not reviewed at either Week 2 or Week 4 were also excluded.
Arm/Group | Lansoprazole
Number analyzed (Participants) | 12653
Age, Customized [Number; unit: participants]
  < 65 years | 6691
  ≥ 65 years | 5962
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7417
  Male | 5236
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 12653
Region of Enrollment [Number; unit: participants]
  Japan | 12653
Body Mass Index (BMI) [Number; unit: participants]
  BMI < 25 kg/m^2 | 6043
  BMI ≥ 25 kg/m^2 and < 30 kg/m^2 | 3083
  BMI ≥ 30 kg/m^2 | 472
  BMI Unknown | 3055
History of Gastroesophageal Reflux Disease [Number; unit: participants]
  Initial | 7128
  Recurrence | 2498
  Unknown | 3027
Duration of Dyspeptic Symptoms [Number; unit: participants]
  < 1 month | 5832
  > 1 month and ≤ 3 months | 3080
  > 3 months and ≤ 6 months | 802
  > 6 months | 1442
  Unknown | 1497
Marked Kyphosis [Number; unit: participants]
  No | 12148
  Yes | 505
Helicobacter pylori (H. pylori) Infection at the Start of Takepron Treatment [Number; unit: participants]
  Negative | 2214
  Positive | 689
  Unknown | 9750

OUTCOME MEASURES:

1. Primary Outcome: Subjective Symptom Improvement Rate
Description: Subjective symptoms were evaluated as "Disappeared," "Improved," "No change," "Worsened," or "Unclear." These categories were based on investigator's definitions. At Week 4, the rate of improvement (i.e. the frequency of an evaluation of "Disappeared" + "Improved") was calculated for each symptom. The percentage of participants with Improvement by symptom was reported.
Time Frame: Start of treatment and Week 4
Population: Efficacy set included all enrolled participants with data available (8 patients were excluded for Investigator's medical reasons; 41 were excluded for other reasons), 1402 patients who did not visit the study site after initial prescription and 861 patients whose questionnaires were not reviewed at either Week 2 or Week 4 were also excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 12653
percentage of participants
  Heartburn | 75.7
  Acid regurgitation | 73.5
  Postorandial fullness | 68.6
  Early satiety | 65.3
  Epigastric pain | 69.1
  Epigastric burning | 73.0
  Upper abdominal bloating | 64.8
  Nausea/vomiting | 66.4
  Belching | 61.6

2. Secondary Outcome: Frequency of Adverse Events (Adverse Drug Reactions)
Description: Adverse events observed during the observation period were collected by symptom. For adverse drug reactions, frequencies were tabulated by type and seriousness. Adverse events were defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with administration of lansoprazole whether or not it was considered related to treatment. Among these, events that were considered as having a causal relationship with lansoprazole were defined as adverse drug reactions. The rate of participants with adverse events (adverse drug reactions) was reported.
Time Frame: 4 Weeks
Population: Safety analysis set included all enrolled participants with data available (8 patients were excluded for Investigator's medical reasons; 41 were excluded for other reasons), 1402 patients who did not visit the study site after initial prescription were also excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 13514
percentage of participants
  Adverse drug reaction(s) | 0.69
  Diarrhoea | 0.16
  Urticaria | 0.08
  Rash | 0.07
  Constipation | 0.04
  Nausea | 0.04
  Abdominal distension | 0.02
  Stomatitis | 0.02
  Dizziness | 0.02
  Dysgeusia | 0.02
  Headache | 0.02
  Drug eruption | 0.02
  Feeling abnormal | 0.01
  Hypoaesthesia | 0.01
  Somnolence | 0.01
  Dyspnoea | 0.01
  Oropharyngeal discomfort | 0.01
  Pruritus | 0.01
  Pruritus generalised | 0.01
  Palpitations | 0.01
  Abdominal pain | 0.01
  Abdominal pain lower | 0.01
  Change of bowel habit | 0.01
  Meteorism | 0.01
  Gastrooesophageal reflux disease | 0.01
  Oral discomfort | 0.01
  Oral mucosal eruption | 0.01
  Abdominal discomfort | 0.01
  Chest pain | 0.01
  Face oedema | 0.01
  Oedema | 0.01
  Thirst | 0.01
  Decreased appetite | 0.01
  Back pain | 0.01
  Sleep disorder | 0.01
  Cough | 0.01
  Acne | 0.01
  Eczema | 0.01
  Erythema multiforme | 0.01
  Toxic skin eruption | 0.01
  Hot flush | 0.01

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: Safety analysis set included all enrolled participants with data available (8 excluded for Investigator's medical reasons; 41 excluded for other reasons), 1402 did not visit site after initial prescription were excluded 1.Serious adverse events; other (not serious) adverse events; 2.Grouped by organ system with number and frequency of events
Arm/Group | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 10/13514
Other Adverse Events (participants affected / at risk) | 0/13514
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lansoprazole (N=13514)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no control groups in this single-arm study. The observed subjective symptom improvement rates and frequency of adverse drug reactions may be used in an exploratory manner to understand drug use but cannot be treated as verified results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.